CLINICAL TRIAL: NCT00171119
Title: A 24-Week Study to Assess Blood Pressure Independent Effects of Valsartan Treatment, Benazepril Treatment and Combination of Both Valsartan and Benazepril Treatment on Urinary Albumin Excretion Rate With Type II Diabetes Mellitus and Microalbuminuria
Brief Title: A Study in Patients With Diabetes Mellitus Type II of the Effect on Albuminuria of 24 Week Treatment With Valsartan, Benazepril, and Valsartan+Benazepril
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489ATR05
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension; Diabetic Nephropathy
Keywords: HYPERTENSION; DIABETES MELLITUS TYPE II; VALSARTAN; BENAZAPRIL
MeSH Terms: conditions — Hypertension; Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
The purpose of this study is to evaluate the efficacy of valsartan, benazepril or the combination of both in reduction of microalbuminuria in Type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged 35-75 years with type 2 diabetes mellitus and recent evidence of persistent microalbuminuria
* patients with a median (of 3 samples) timed overnight UAER in the microalbuminuric range of 20-200 g/min in the formal screening period prior to entry
* patients who give written, signed, informed consent.
* patients with/without mild /moderate hypertension.
* patients who are not on hypertensive treatment, or if they are already on treatment, those who accept to enter a 3 weeks no-treatment wash-out period before switching their treatment.
* patients without any accompanying systemic disease

Exclusion Criteria:

* pregnant or nursing women, or women of childbearing potential not using an acceptable method of contraception
* patients with type I diabetes mellitus defined by onset below the age of 35 years and requiring insulin within the first year after diagnosis

Other protocol-defined exclusion criteria may apply.

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine albumin excretion rate after 24 weeks

SECONDARY OUTCOMES:
Change from baseline in urine albumin excretion rate after 24 weeks in those patients with blood pressure greater than 140/90, or who had previously taken blood pressure medicine, at study entry
Percent of patients returning to normal urine albumin excretion rate after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland